CLINICAL TRIAL: NCT02411591
Title: A Single-Arm, Multicenter, Phase 1b Study With an Expansion Cohort to Evaluate Safety and Efficacy of Necitumumab in Combination With Abemaciclib in Treatment of Patients With Stage IV Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of Necitumumab and Abemaciclib in Participants With Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 15573; I4X-MC-JFCU (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-03-17; First posted 2015-04-08 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2019-07-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — necitumumab; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Necitumumab + Abemaciclib (Experimental): Cohort 1 Part A: Necitumumab 800 mg administered intravenously (IV) on Days 1 and 8, followed by abemaciclib 100 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
  Cohort 2 Part A: Necitumumab 800 mg administered IV on Days 1 and 8, followed by abemaciclib 150 mg given orally every 12 hours on Days 1 to 21. Treatment may continue until discontinuation criterion is met.
  Cohort 3 Part A: Necitumumab 800 mg administered IV on Days 1 and 8, followed by abemaciclib 200 mg given orally every 12 hours on Days 1 to 21. Treatment may continue until discontinuation criterion is met.
  Part B (expansion cohort): Necitumumab 800 mg administered IV on Days 1 and 8, followed by abemaciclib 150 mg given orally every 12 hours on Days 1 to 21. Treatment may continue until discontinuation criterion is met.
  Interventions: Drug: Necitumumab; Drug: Abemaciclib

INTERVENTIONS:
Drug: Necitumumab — Administered IV.
  Other Names: LY3012211
Drug: Abemaciclib — Administered orally.
  Other Names: LY2835219

SUMMARY:
This is medical research evaluating the safety and efficacy of two new medicines (necitumumab and abemaciclib), administered in combination in participants affected by a defined type of advanced lung cancer (stage IV non-small-cell lung cancer).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC Stage IV:

  * Part A: NSCLC Stage IV (any type).
  * Part B: NSCLC Stage IV (squamous and nonsquamous).
* Measurable disease at the time of study entry as defined by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1).
* The participant must have progressed after platinum-based chemotherapy AND have received a maximum of 1 other prior chemotherapy for advanced and/or metastatic disease OR must be judged by the physician as ineligible for further standard second-line chemotherapy. Prior treatment with epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI) and anaplastic lymphoma kinase (ALK) inhibitors is mandatory in participants whose tumor has EGFR-activating mutations or ALK translocations. Prior targeting agents and neoadjuvant/adjuvant therapies are permitted with the exception of cyclin-dependent kinase (CDK)4/6-targeting agents or necitumumab.
* The participant has tumor tissue available for biomarker analyses.
* The participant has an Eastern Cooperative Oncology Group performance status score of 0-1.
* Have adequate organ functions.

Exclusion Criteria:

* The participant is currently enrolled in a clinical trial involving an investigational product or non-approved use of a drug or device. Prior treatment with cyclin-dependent kinase 4 and 6 (CDK4/6) - targeting agents or necitumumab is not permitted.
* Have a serious concomitant systemic disorder or significant cardiac disease.
* The participant has undergone major surgery or received any investigational therapy in the 30-days prior to study enrollment.
* The participant has undergone chest irradiation within 4 weeks prior to receiving study treatment.
* The participant has brain metastases that are symptomatic.
* History of arterial or venous thromboembolism within 3 months prior to study enrollment. Participants with a history of venous thromboembolism beyond 3 months prior to study enrollment can be enrolled if they are appropriately treated with low molecular weight heparin.
* The participant has active infection requiring systemic therapy.
* The participant has a known allergy / history of hypersensitivity reaction to any of the treatment components, including any ingredient used in the formulation of necitumumab or abemaciclib, or any other contraindication to one of the administered treatments.
* The participant is pregnant or breastfeeding.
* The participant has a concurrent active malignancy. Previous history of malignancy is permitted, provided that the participant has been free of disease for ≥3 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, preinvasive carcinoma of the cervix, or any cancers that in the judgment of the investigator and sponsor may not affect the interpretation of results (for example, prostate, bladder).
* History of interstitial lung disease or an active non-infectious pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2019-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- Belgium (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Charleroi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Leuven
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Roeselare
- France (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Brest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Bron
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Pau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Strasbourg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), or speak with your personal physician., Villejuif
- Spain (3):
  - Hospital Universitario Ramon y Cajal, Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Click here for more information about this study: A Study of Necitumumab (LY3012211) and Abemaciclib (LY2835219) in Participants With Stage IV Non-small Cell Lung Cancer (NSCLC) — https://www.lillytrialguide.com/en-US/studies/non-small-cell-lung-cancer/JFCU#?postal=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study has 2 parts (Part A and Part B). Part A is a dose-escalation study to determine the recommended dose of abemaciclib in combination with necitumumab Part B (expansion cohort). Completers completed the 2 cycles, with required assessment, had progressive disease or died due to any cause, alive and on study at conclusion but off treatment.
Groups:
- Cohort 1 (Necitumumab 800 mg + Abemaciclib 100 mg): Part A: Necitumumab 800 milligram (mg) was administered intravenously (IV) on Days 1 and 8, followed by abemaciclib 100 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
- Cohort 2 (Necitumumab 800 mg + Abemaciclib 150 mg): Part A: Necitumumab 800 mg administered IV on Days 1 and 8, followed by abemaciclib 150 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
  Part B: (expansion cohort): Necitumumab 800 mg administered IV on Days 1 and 8, followed by abemaciclib 150 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
- Cohort 3 (Necitumumab 800 mg + Abemaciclib 200 mg): Part A: Necitumumab 800 mg was administered IV on Days 1 and 8, followed by abemaciclib 200 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
Period: Overall Study
Arm/Group | Cohort 1 (Necitumumab 800 mg + Abemaciclib 100 mg) | Cohort 2 (Necitumumab 800 mg + Abemaciclib 150 mg) | Cohort 3 (Necitumumab 800 mg + Abemaciclib 200 mg)
Started | 3 | 57 | 6
Part A | 3 | 6 | 6
Expansion Cohort Part B | 0 | 51 | 0
Progressive Disease | 3 | 42 | 3
Death | 0 | 2 | 0
Completed | 3 | 47 | 3
Not Completed | 0 | 10 | 3
Not completed — Adverse Event | 0 | 4 | 2
Not completed — Withdrawal by Subject | 0 | 3 | 0
Not completed — Physician Decision | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study drug. Cohort 2 includes total number of participants in Part A and evaluable participants of Part B.
Groups:
- Cohort 1 (Necitumumab 800 mg + Abemaciclib 100 mg): Part A: Necitumumab 800 mg was administered IV on Days 1 and 8, followed by abemaciclib 100 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
- Cohort 2 (Necitumumab 800 mg + Abemaciclib 150 mg): Part A: Necitumumab administered intravenously (IV) on Days 1 and 8, followed by abemaciclib given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
  Part B (expansion cohort) : Necitumumab administered IV on Days 1 and 8, followed by abemaciclib given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
- Cohort 3 (Necitumumab 800 mg + Abemaciclib 200 mg): Part A: Necitumumab 800 mg was administered IV on Days 1 and 8, followed by abemaciclib 200 mg given orally Q12H on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Necitumumab 800 mg + Abemaciclib 100 mg) | Cohort 2 (Necitumumab 800 mg + Abemaciclib 150 mg) | Cohort 3 (Necitumumab 800 mg + Abemaciclib 200 mg) | Total
Number analyzed (Participants) | 3 | 57 | 6 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.33 (2.31) | 61.42 (10.58) | 49.00 (7.59) | 60.33 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 17 | 1 | 19
  Male | 2 | 40 | 5 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 1 | 13 | 1 | 15
  Unknown or Not Reported | 2 | 42 | 5 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 16 | 1 | 18
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 41 | 5 | 48
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 1 | 9 | 1 | 11
  France | 2 | 45 | 5 | 52
  Spain | 0 | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Abemaciclib Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as one of the following adverse events (AEs), occurring in Cycle 1 if considered to be definitely, probably, or possibly related to necitumumab and abemaciclib: Grade 3 or 4 nonhematologic toxicity according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI-CTCAE v4.0), except for nausea, vomiting, diarrhea, or electrolyte disturbance. Grade 3 or 4 nausea, vomiting, or diarrhea that persists more than 2 days despite maximal supportive intervention. Grade 3 thrombocytopenia with bleeding requiring transfusion. Grade 4 thrombocytopenia with or without bleeding. Grade 4 neutropenia that persists more than 5 days.
Time Frame: Baseline through Cycle 1 (Up to 21 Days)
Population: All participants who received at least one dose of study drug and had evaluable DLTs.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2 (Necitumumab 800 mg + Abemaciclib 150 mg): Part A: Necitumumab 800 mg was administered IV on Days 1 and 8, followed by abemaciclib 150 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
- Cohort 3 (Necitumamab 800 mg + Abemaciclib 200 mg): Part A: Necitumumab 800 mg was administered IV on Days 1 and 8, followed by abemaciclib 200 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
Arm/Group | Cohort 1 (Necitumumab 800 mg + Abemaciclib 100 mg) | Cohort 2 (Necitumumab 800 mg + Abemaciclib 150 mg) | Cohort 3 (Necitumamab 800 mg + Abemaciclib 200 mg)
Number analyzed (Participants) | 3 | 6 | 6
Participants | 0 | 1 | 3

2. Primary Outcome: Progression Free Survival (PFS) Rate at 3 Months (Percentage of Participants With PFS at 3 Months)
Description: PFS is defined as the time from baseline until first observation of progressive disease(PD) defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause.PD was at least 20% increase in sum of diameters of target lesions with reference being smallest sum on study and an absolute increase of at least 5 millimeter (mm) or unequivocal progression of non-target lesions,or 1 or more new lesions.If participant does not have complete baseline disease assessment,PFS time censored at date of randomization, regardless of whether or not objectively determined disease progression or death observed for participant.If participant was not known to have died or have objective progression as of data inclusion cutoff date for analysis, the PFS time censored at last adequate tumor assessment date.The use of new anticancer therapy prior to occurrence of PD resulted in censoring at the date of last radiographic assessment prior to initiation of new therapy.
Time Frame: Baseline to measured progressive disease or death due to any cause (3 Months)
Population: All enrolled participants who received at least one dose of study drug and had evaluable PFS data. Cohort 2 number of censored participants is 10. Cohort 2 includes total number of participants in Part A and evaluable participants of Part B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 2 (Necitumumab 800 mg + Abemaciclib 150 mg): Part A: Necitumumab 800 mg was administered IV on Days 1 and 8, followed by abemaciclib 150 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
  Part B (expansion cohort): Necitumumab 800 mg administered IV on Days 1 and 8, followed by abemaciclib 150 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
Arm/Group | Cohort 1 (Necitumumab 800 mg + Abemaciclib 100 mg) | Cohort 2 (Necitumumab 800 mg + Abemaciclib 150 mg) | Cohort 3 (Necitumumab 800 mg + Abemaciclib 200 mg)
Number analyzed (Participants) | 3 | 57 | 6
percentage of participants | 66.7 [5.4 to 94.5] | 32.3 [20.4 to 44.8] | 50.0 [11.1 to 80.4]

3. Secondary Outcome: Percentage of Participants Who Achieve Best Overall Tumor Response of Complete or Partial Response (Objective Response Rate [ORR])
Description: ORR was the percentage of participants achieving a best overall response of complete response (CR) or partial response (PR) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions (taking as reference the baseline sum LD), no progression of nontarget lesions, and no appearance of new lesions. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. Confidence intervals are based on Clopper-Pearson method.
Time Frame: Baseline to measured progressive disease or start of new anti-cancer therapy (up to 21 months)
Population: All enrolled participants who received at least one dose of study drug and had evaluable ORR data in cohorts 1, 2 and 3. Cohort 2 includes total number of participants in Part A and evaluable participants of Part B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 2 (Necitumumab 800 mg + Abemaciclib 150 mg): Part A: Necitumumab 800 mg administered intravenously (IV) on Days 1 and 8, followed by abemaciclib 150 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
  Part B (expansion cohort): Necitumumab 800 mg administered IV on Days 1 and 8, followed by abemaciclib 150 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
- Total Enrolled Participants (Necitumumab + Abemaciclib): Cohorts 1, 2 and 3 combined. Necitumumab 800 mg was administered IV on Days 1 and 8, followed by abemaciclib 100 mg, 150 mg or 200 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
Arm/Group | Cohort 1 (Necitumumab 800 mg + Abemaciclib 100 mg) | Cohort 2 (Necitumumab 800 mg + Abemaciclib 150 mg) | Cohort 3 (Necitumumab 800 mg + Abemaciclib 200 mg) | Total Enrolled Participants (Necitumumab + Abemaciclib)
Number analyzed (Participants) | 3 | 57 | 6 | 66
percentage of participants
  Overall Response Rate | 66.7 [9.4 to 99.2] | 5.3 [1.1 to 14.6] | 0.0 [0.0 to 45.9] | 7.6 [2.5 to 16.8]
  PR | 66.7 [9.4 to 99.2] | 5.3 [1.1 to 14.6] | 0.0 [0.0 to 45.9] | 7.6 [2.5 to 16.8]
  SD | 33.3 [0.8 to 90.6] | 42.1 [29.1 to 55.9] | 66.7 [22.3 to 95.7] | 43.9 [31.7 to 56.7]
  PD | 0.0 [0.0 to 70.8] | 47.4 [34.0 to 61.0] | 16.7 [0.4 to 64.1] | 42.4 [30.3 to 55.2]

4. Secondary Outcome: Pharmacokinetics (PK): Predose Concentration (Cmin) of Necitumumab
Description: Predose necitumumab concentration data following doses of 800 mg administered Day 1 and 8 of a 3-week cycle as an intravenous (IV) infusion over 60 minutes.
Time Frame: Cycle 1, Day 8 (C1D8) and C2,3,5,7 D1: Predose
Population: All participants who received same dose of necitumumab, pre-specified to assess as single group and had evaluable PK data.
Measure: Geometric Mean (Standard Deviation); unit: microgram/milliliter (μg/mL)
Groups:
- Necitumumab: Necitumumab 800 mg was administered IV on Days 1 and 8, of a 3-week cycle.
Arm/Group | Necitumumab
Number analyzed (Participants) | 61
microgram/milliliter (μg/mL)
  Cycle 1, Day 8 | 64.1 (43.1)
  Cycle 2, Day 1 | 49.6 (63.8)
  Cycle 3, Day 1 | 93.8 (44.1)
  Cycle 5, Day 1 | 160 (50.3)
  Cycle 7, Day 1 | 165 (42.1)

5. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Necitumumab
Description: Maximum necitumumab concentration data following doses of 800 mg administered Day 1 and 8 of a 3-week cycle as an intravenous (IV) infusion over 60 minutes.
Time Frame: Cycle 1, Day 1 (C1D1): 0.25, 2,4,10 hours(h) post dose, C1D8: 0.25h post dose, Cycle 2, Day 1 (C2D1): 0.25, 2,4,10h post dose; C3,5,7 D1: 0.25h post dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Necitumumab
Number analyzed (Participants) | 61
μg/mL
  Cycle 1, Day 1 | 228 (45.6)
  Cycle 1, Day 8 (D8) | 304 (21.9)
  Cycle 2, Day 1 | 270 (25.6)
  Cycle 3, Day 1 | 318 (43.7)
  Cycle 5, Day 1 | 356 (42.7)
  Cycle 7, Day 1 | 350 (24.7)

6. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Abemaciclib
Description: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Abemaciclib summary of LSN3106729 noncompartmental PK parameters after twice daily oral dose of Abemaciclib.
Time Frame: Cycle 1, Day 1 (C1D1): 0.25, 2,4,6,8,10 hours(h) post dose, C1D8: 0.25h post dose, C2D1: 0.25, 2,4,6,8,10h post dose; C3,5,7 D1: 0.25h post dose
Population: All participants who received at least one dose of abemaciclib and had evaluable PK data for Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Groups:
- Abemaciclib 100 mg: Necitumumab 800 mg administered IV on Days 1 and 8 followed by abemaciclib 100 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
- Abemaciclib 150 mg: Necitumumab 800 mg administered IV on Days 1 and 8 followed by abemaciclib 150 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
- Abemaciclib 200 mg: Necitumumab 800 mg administered IV on Days 1 and 8 followed by abemaciclib 200 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
Arm/Group | Abemaciclib 100 mg | Abemaciclib 150 mg | Abemaciclib 200 mg
Number analyzed (Participants) | 3 | 5 | 5
nanogram/milliliter (ng/mL) | 15.6 (146) | 26 (148) | 38.2 (80)

7. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) From Zero to the Last Time Point (AUC[0-tlast]) Abemaciclib
Description: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) From Zero to the Last Time Point (AUC[0-tlast]) summary of LSN3106729 noncompartmental PK parameters after twice daily oral dose of Abemaciclib. (tlast = 10 hours)
Time Frame: Cycle 1, Day 1 (C1D1): 0.25, 2,4,6,8,10 hours(h) post dose
Population: All participants who received at least one dose of abemaciclib and had evaluable PK data for Part A.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter (hr*ng/mL)
Arm/Group | Abemaciclib 100 mg | Abemaciclib 150 mg | Abemaciclib 200 mg
Number analyzed (Participants) | 3 | 5 | 5
hour*nanogram/milliliter (hr*ng/mL) | 118 (200) | 209 (136) | 336 (83)

8. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR), Partial Response (PR), and Stable Disease (SD) (Disease Control Rate [DCR])
Description: Disease Control Rate (DCR) is defined as the percentage of participants achieving a best overall response of stable disease (SD), PR, or CR. DCR used the same denominator as defined in ORR. Among participants counted in the denominator, the numerator counted those with a confirmed best tumor response of SD, PR, or CR per RECIST v1.1. Confidence intervals are based on Clopper-Pearson method.
Time Frame: Baseline to measured progressive disease or start of new anti-cancer therapy (up to 21 months)
Population: All enrolled participants who received at least one dose of study drug and had evaluable ORR data in cohorts 1, 2 and 3.Cohort 2 includes total number of participants in Part A and evaluable participants of Part B.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 (Necitumumab 800 mg + Abemaciclib 100 mg) | Cohort 2 (Necitumumab 800 mg + Abemaciclib 150 mg) | Cohort 3 (Necitumumab 800 mg + Abemaciclib 200 mg) | Total Enrolled Participants (Necitumumab + Abemaciclib)
Number analyzed (Participants) | 3 | 57 | 6 | 66
percentage of participants | 100 [29.2 to 100.0] | 47.4 [34.0 to 61.0] | 66.7 [22.3 to 95.7] | 51.5 [38.9 to 64.0]

9. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from the date of study enrollment to the date of death from any cause. For each participant who is not known to have died as of the data -inclusion cutoff date for a particular analysis, OS was censored for that analysis at the last known alive date.
Time Frame: Baseline to date of death from any cause (24 Months)
Population: All enrolled participants who received at least one dose of study drug and had evaluable overall survival (OS) data. Cohort 2 includes total number of participants in Part A and evaluable participants of Part B. Participants censored in cohort 1 = 2, cohort 2 = 1 and cohort 3 = 21.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 (Necitumumab 800 mg + Abemaciclib 100 mg) | Cohort 2 (Necitumumab 800 mg + Abemaciclib 150 mg) | Cohort 3 (Necitumumab 800 mg + Abemaciclib 200 mg)
Number analyzed (Participants) | 3 | 57 | 6
Months | NA [18.20 to NA] — 95% Confidence Interval (CI) had not matured yet and median was not calculable. | 6.93 [4.96 to 12.85] | 13.45 [1.31 to 18.53]

ADVERSE EVENTS:
Time Frame: Up to 21 Months
Description: All enrolled participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Necitumumab 800 mg + Abemaciclib 100 mg: Necitumumab 800 mg was administered IV on Days 1 and 8, followed by abemaciclib 100 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
- Necitumumab 800 mg + Abemaciclib 150 mg: Necitumumab 800 mg administered intravenously (IV) on Days 1 and 8, followed by abemaciclib 150 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
- Necitumumab 800 mg + Abemaciclib 200 mg: Necitumumab 800 mg was administered IV on Days 1 and 8, followed by abemaciclib 200 mg given orally every 12 hours on Days 1 to 21. (21 day cycles.) Treatment may continue until discontinuation criterion is met.
Arm/Group | Necitumumab 800 mg + Abemaciclib 100 mg | Necitumumab 800 mg + Abemaciclib 150 mg | Necitumumab 800 mg + Abemaciclib 200 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 5/57 | 2/6
Serious Adverse Events (participants affected / at risk) | 2/3 | 25/57 | 4/6
Other Adverse Events (participants affected / at risk) | 3/3 | 57/57 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Necitumumab 800 mg + Abemaciclib 100 mg (N=3) | Necitumumab 800 mg + Abemaciclib 150 mg (N=57) | Necitumumab 800 mg + Abemaciclib 200 mg (N=6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 5 (6) | 0 (0)
Fatigue (General disorders) | 0 (0) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 1 (1)
Vascular stent thrombosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Necitumumab 800 mg + Abemaciclib 100 mg (N=3) | Necitumumab 800 mg + Abemaciclib 150 mg (N=57) | Necitumumab 800 mg + Abemaciclib 200 mg (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 21 (45) | 3 (4)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (9) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 2 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 7 (7) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 8 (8) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 29 (49) | 3 (6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 24 (32) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 7 (8) | 3 (5)
Tooth discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 16 (24) | 3 (4)
Asthenia (General disorders) | 1 (1) | 8 (12) | 1 (1)
Fatigue (General disorders) | 2 (6) | 29 (49) | 3 (4)
General physical health deterioration (General disorders) | 0 (0) | 4 (4) | 0 (0)
Mucosal dryness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 3 (3) | 1 (1)
Pain (General disorders) | 0 (0) | 5 (5) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 10 (10) | 2 (2)
Xerosis (General disorders) | 1 (1) | 4 (4) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 4 (5) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 5 (5) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 5 (8) | 1 (1)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 2 (3) | 6 (9) | 3 (3)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 5 (6) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (4) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 13 (23) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 9 (18) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 11 (28) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 7 (9) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 21 (24) | 4 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 12 (17) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 20 (29) | 1 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 4 (7) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 8 (18) | 1 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 5 (5) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 6 (6) | 3 (3)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 5 (5) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0/1 (0) | 1/17 (1) | 0/1 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 10 (10) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 21 (21) | 1 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (6) | 26 (41) | 3 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (3) | 15 (20) | 4 (4)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (9) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (7) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 8 (23) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-05-12): https://cdn.clinicaltrials.gov/large-docs/91/NCT02411591/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT02411591/SAP_001.pdf